CLINICAL TRIAL: NCT05793125
Title: Correlation Between Pulmonary Artery Doppler And Neonatal Outcome In Hypertensive Disorders Of Pregnancy
Brief Title: Pulmonary Artery Doppler And Neonatal Outcome In Hypertensive Disorders Of Pregnancy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran Amin, assistant lecturer of Obstetrics and Gynecology, Cairo University
Other Study IDs: Pregnancy induced hypertension
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography — A full obstetrics ultrasound scan will be performed within 24 hours before delivery to document fetal biometry, estimated fetal weight and correlate it to fetal growth charts to exclude IUGR, amniotic fluid index and umbilical artery Doppler studies.
  Fetal echocardiography will be done.Pulmonary artery Doppler ﬂow waveforms, including pulsatility index, resistance index, systolic-to-diastolic ratio, peak systolic velocity, and acceleration time to ejection time (At/Et) ratio will be measured in the main pulmonary artery.

SUMMARY:
To correlate fetal Pulmonary artery Doppler parameters with neonatal outcome in patients diagnosed with hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
Hypertensive disorders include gestational hypertension, preeclampsia, chronic hypertension, preeclampsia superimposed on chronic hypertension. They complicate up to 10% of pregnancies. As a group they are one member of the deadly triad, along with hemorrhage and infection, that contributes greatly to maternal morbidity.

Preeclampsia, either alone or superimposed on chronic hypertension, is the most dangerous. Most hypertension related deaths are preventable. Also, nonsevere preeclampsia may progress rapidly to severe disease causing headache or visual disturbance that precede eclampsia. They also cause epigastic or right upper quadrant pain and elevated hepatic transaminases that frequently accompany hepatocellular necrosis, ischemia and edema, thrombocytopenia that represents platelet activation and aggregation, microangiopathic hemolysis, renal involvement and placental abruption. On the long term, preeclampsia is also associated with adverse health problems including chronic hypertension, ischemic heart disease, atherosclerosis, cardiomyopathy, peripheral vascular disease, type 2 diabetes, dyslipidemia, obesity and metabolic syndrome.

Termination of pregnancy is the only known cure for preeclampsia. Moreover, expectant management of preterm severe preeclampsia leads to disastrous results as increase in perinatal mortality rate, placental abruption, eclampsia, renal failure, hypertensive encephalopathy, intracranial hemorrhage or even rupture in hepatic hematoma.

Early attempts have been made to predict fetal maturity on the basis antenatal ultrasonographic parameters including lung characteristics, bowel pattern, placental grading, the presence or absence of intraamniotic particles (vernix caseosa) and the epiphyseal ossification centers appearance and enlargement.

More recently, fetal pulmonary artery Doppler has been used to predict neonatal respiratory rate (RDS). It was found that an elevated acceleration-to-ejection time ratio was significantly associated with neonatal RDS. However such indices cannot be generalized in all cases, especially those with hypertensive disorders of pregnancy who have abnormal trophoblastic invasion of uterine vessels affecting fetoplacental circulation resistance.

To the best of our knowledge, no available studies have correlated fetal pulmonary artery Doppler indices with neonatal outcomes in patients with hypertensive disorders of pregnancy. Presence of such signs of maturity can aid the obstetrician to choose the most appropriate timing for termination especially in low income countries who have limited access to neonatal intensive care units. Being cost effective and non invasive ultrasonography is used as a routine obstetrics scanning tool. This study will help determine the utility of ultrasound and Doppler in assessing the fetal lung maturity in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-42 years old
* Patients who will be diagnosed with hypertensive disorders of pregnancy preoperatively according to (ACOG 2020)
* Those who will undergo elective or emergency termination of pregnancy whether by vaginal or cesarean delivery .
* Primi or multigravida
* With gestational age: 28 0/7 - 37 6/7 weeks

Exclusion Criteria:

* Multifetal pregnancy
* Intrauterine fetal death
* Intrauterine growth restriction (IUGR) which is defined as a rate of fetal growth that is less than normal for the growth potential of that specific infant
* Placental abruption whether diagnosed before or during delivery.
* Absent or reversed umbilical artery end diastolic flow.
* Diabetes with pregnancy either gestational or overt which is defined as any degree of glucose intolerance with an onset or first recognition during pregnancy
* Premature or prelabor rupture of membranes
* BMI above 40 due to technical difficulties to obtain accurate measures
* Major congenital fetal anomalies whether diagnosed before or after delivery
* Maternal fever more than 37.4 degree
* Emergent cases presenting with fetal distress (bradycardia will be defined as fetal heart rate < 110 beat per minute)
* Patient receiving general anesthesia if termination was by cesarean delivery
* Patients receiving narcotics 4 hours before delivery
* Patients with unreliable dates or no crown rump length at first trimester.

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant patients diagnosed with hypertensive disorders undergoing elective or emergency termination of pregnancy in Kasr Alainy hospital.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Acceleration time to ejection time ratio (At/Et) of fetal pulmonary artery Doppler in neonates needing respiratory support | Baseline
  (At/Et) ratio will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome

SECONDARY OUTCOMES:
The pulsatility index (PI) of fetal pulmonary artery Doppler in neonates needing respiratory support | Baseline
  The PI will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome
The resistance index (RI) of fetal pulmonary artery Doppler in neonates needing respiratory support | baseline
  The RI will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome
The systolic to diastolic ratio (S/D) of fetal pulmonary artery Doppler in neonates needing respiratory support | baseline
  The S/D ratio will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome
The peak systolic velocity (PSV) of fetal pulmonary artery Doppler in neonates needing respiratory support | baseline
  The PSV will be measured in the fetal main pulmonary artery Doppler and will be correlated with the neonatal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H El Sawaf, MD, Study Director — Cairo University; Ahmed M Salah, MD, Study Chair — Cairo University
Locations (1):
- Kasralainy Cairo University, Giza, Egypt

REFERENCES:
- [Background] Judy AE, McCain CL, Lawton ES, Morton CH, Main EK, Druzin ML. Systolic Hypertension, Preeclampsia-Related Mortality, and Stroke in California. Obstet Gynecol. 2019 Jun;133(6):1151-1159. doi: 10.1097/AOG.0000000000003290. PMID 31135728
- [Background] Buchanan TA, Xiang AH. Gestational diabetes mellitus. J Clin Invest. 2005 Mar;115(3):485-91. doi: 10.1172/JCI24531. PMID 15765129
- [Background] Churchill D, Duley L, Thornton JG, Moussa M, Ali HS, Walker KF. Interventionist versus expectant care for severe pre-eclampsia between 24 and 34 weeks' gestation. Cochrane Database Syst Rev. 2018 Oct 5;10(10):CD003106. doi: 10.1002/14651858.CD003106.pub3. PMID 30289565
- [Background] Hornberger LK, Sahn DJ. Rhythm abnormalities of the fetus. Heart. 2007 Oct;93(10):1294-300. doi: 10.1136/hrt.2005.069369. No abstract available. PMID 17890709
- [Background] Katsuragi S, Tanaka H, Hasegawa J, Nakamura M, Kanayama N, Nakata M, Murakoshi T, Yoshimatsu J, Osato K, Tanaka K, Sekizawa A, Ishiwata I, Ikeda T; Maternal Death Exploratory Committee in Japan and Japan Association of Obstetricians and Gynecologists. Analysis of preventability of hypertensive disorder in pregnancy-related maternal death using the nationwide registration system of maternal deaths in Japan. J Matern Fetal Neonatal Med. 2019 Oct;32(20):3420-3426. doi: 10.1080/14767058.2018.1465549. Epub 2018 Apr 26. PMID 29699420
- [Background] Mahony BS, Bowie JD, Killam AP, Kay HH, Cooper C. Epiphyseal ossification centers in the assessment of fetal maturity: sonographic correlation with the amniocentesis lung profile. Radiology. 1986 May;159(2):521-4. doi: 10.1148/radiology.159.2.3515425.
- [Background] McCowan LM, Figueras F, Anderson NH. Evidence-based national guidelines for the management of suspected fetal growth restriction: comparison, consensus, and controversy. Am J Obstet Gynecol. 2018 Feb;218(2S):S855-S868. doi: 10.1016/j.ajog.2017.12.004. PMID 29422214
- [Background] Wang YX, Arvizu M, Rich-Edwards JW, Wang L, Rosner B, Stuart JJ, Rexrode KM, Chavarro JE. Hypertensive Disorders of Pregnancy and Subsequent Risk of Premature Mortality. J Am Coll Cardiol. 2021 Mar 16;77(10):1302-1312. doi: 10.1016/j.jacc.2021.01.018. PMID 33706872
- [Background] Varner S, Sherman C, Lewis D, Owens S, Bodie F, McCathran CE, Holliday N. Amniocentesis for fetal lung maturity: will it become obsolete? Rev Obstet Gynecol. 2013;6(3-4):126-34. PMID 24826202
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin Summary, Number 222. Obstet Gynecol. 2020 Jun;135(6):1492-1495. doi: 10.1097/AOG.0000000000003892. PMID 32443077